CLINICAL TRIAL: NCT01599078
Title: Local Delivery of Paclitaxel Via the TAPAS Catheter to Prevent Restenosis From Percutaneous Femoropopliteal Intervention (PacTAP Study): A Double Blind, Randomized Control Study
Brief Title: Local Delivery of Paclitaxel Via the TAPAS Catheter to Prevent Restenosis From Percutaneous Femoropopliteal Intervention
Acronym: PacTAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Midwest Cardiovascular Research Foundation (Other)
Collaborators: Spectranetics Corporation (Industry)
Responsible Party: Principal Investigator, Eric J Dippel, MD, President, Midwest Cardiovascular Foundation, Midwest Cardiovascular Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCRF-001-EJD
Record Dates: First submitted 2012-05-13; First posted 2012-05-15 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Restenosis; Peripheral Arterial Disease
Keywords: Restenosis; Angioplasty; Stent; Atherectomy; Femoral Artery; Popliteal Artery; Paclitaxel
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Paclitaxel (Active Comparator)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Drug dosing is 3mcg/mm3 of artery treated with percutaneous revascularization. Drug will be administered via the TAPAS catheter and allowed to dwell for 5 minutes.
  Other Names: Taxol
  Arms: Paclitaxel
Drug: Placebo — Saline will be administered intra-arterially via the TAPAS catheter following percutaneous revascularization. The dwell time will be 5minutes.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of administering intra-arterial paclitaxel in the femoropopliteal arteries via the TAPAS catheter following percutaneous revascularization to prevent restenosis.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) of the lower extremities is an extremely prevalent disorder and is an important cause of morbidity that affects more than 10 million people in the United States. This disorder is typically caused by atherosclerosis that limits blood flow to the limbs, particularly due to stenosis or occlusion of the superficial femoral artery (SFA) and/or popliteal artery. Although many patients are asymptomatic or are treated with lifestyle changes, such as exercise therapy, or pharmacological treatment, including statins and anti-platelet therapy, about 10-15% of patients have progressive symptoms which in severe cases may lead to amputation.

Endovascular treatment with percutaneous vascular intervention (PVI), which includes percutaneous transluminal angioplasty (PTA), stenting, atherectomy and thrombolytic therapy, can provide excellent acute success rates greater than 90-95% However, the intermediate to long-term patency rates of these arteries is hampered by neointimal hyperplasia resulting in restenosis of the artery. This occurs with all endovascular therapy to some degree in both the coronary and peripheral arena. With PVI in the superficial femoral and popliteal arteries the restenosis rates are approximately 30-40% at 12 months, depending on the complexity and severity of the disease.

In the coronary field, stents are now coated with anti-restenotic pharmacologic agents (drug eluting stents-DES) such as paclitaxel and sirolimus-like drugs that prevent neointimal growth. There have been published reports of significant efficacy in preventing restenosis in the SFA by coating balloons with paclitaxel (drug eluting balloons-DEB) as well as a nitinol stent. Despite the fact that these products are CE Mark approved and available in Europe, currently there are no US FDA approved drug-eluting devices for use in PVI. Thus, there remains a need for an alternative therapy to prevent restenosis in the SFA following endovascular intervention.

Administration of intra-arterial paclitaxel mixed with iodinated contrast has been shown to inhibit restenosis in a porcine coronary model.

Delivering paclitaxel intra-arterially in the coronary tree following stent implantation has shown benefit in reducing the incidence of restenosis. The novel Targeted Adjustable Pharmaceutical Application System (TAPAS)-TAPAS Catheter Therapeutic Infusion System (ThermopeutiX, San Diego, CA, USA)-is a drug delivery catheter that consists of a proximal and distal occlusion balloon with an adjustable length that allows a drug to dwell in a specific segment of the artery for a period of time. The drug can then be aspirated and discarded to avoid systemic exposure.

The PacTAP study is a randomized, double blind, placebo-control study to assess the safety and efficacy of delivering intra-arterial paclitaxel via the TAPAS catheter following PVI to prevent restenosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Subject able to provide informed consent and agree to all follow up requirements.
* Peripheral arterial disease with Rutherford Class 2-5.
* Successful percutaneous revascularization of the femoropopliteal artery (< 20% residual stenosis by visual estimate) using standard techniques per discretion of the local operator.
* The femoropopliteal Reference Vessel Diameter (RVD) must be ≥4.0 mm and ≤7.0 mm

Exclusion Criteria:

* Patient is pregnant or breast feeding. (Female subjects of childbearing potential must have negative serum pregnancy test the day of the procedure.)
* Life expectancy < 12 months.
* Contraindication to aspirin, anti-platelet/anti-coagulant therapies required for procedure/follow up.
* Known allergy to contrast media that cannot adequately be pre-medicated prior to study procedure.
* Known allergy to paclitaxel.
* Uncontrolled hypercoagulability or history of HIT or HITTS syndrome.
* Simultaneous enrollment in another investigational device or drug study.
* Previous intervention of the target limb with a drug eluting stent or drug eluting balloon.
* Absence of at least 1 TIMI-3 vessel run off into the foot.
* Total bilirubin > 2x upper limit of normal (ULN).
* ALT or AST > 3x ULN.
* Platelet count < 100,000/mm3.
* White blood cell count < 1.5/mm3.
* Any evidence of perforation or dye extravasation during the index procedure, even if successfully treated with a covered stent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Primary Patency | 6 months
  Loss of primary patency will occur for any clinically driven Target Lesion Revascularization (TLR) or a Peak Systolic Velocity Ratio (PSVR) of > 2.5 on Duplex Ultrasound (DUS)
Primary Safety | 30 days
  Freedom from death, major amputation in the target limb, or Target Lesion Revascularization (either surgical or endovascular)

SECONDARY OUTCOMES:
Primary Patency at 12 months | 12 months
  Loss of primary patency will occur for any clinically driven Target Lesion Revascularization (TLR) or a Peak Systolic Velocity Ratio (PSVR) of > 2.5 on Duplex Ultrasound (DUS)
Primary Assisted Patency | 6 and 12 months
  Patency of the target vessel regardless of secondary interventions performed to restore blood flow after restenosis.
Secondary Patency | 6 and 12 months
  Patency of the target vessel regardless of secondary interventions performed to restore blood flow after reocclusion.
Functional Status | 30 days, 6 months, and 12 months
  Walking Impairment Questionnaire (WIQ), and Rutherford Classification.
Secondary Safety | 30 days, 6 months, and 12 months
  Any adverse events associated with the use of paclitaxel, such as, but not limited to: hypotension, anaphylactic reactions, nausea, vomiting, diarrhea, pancytopenia, neuropathy, alopecia.

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Dippel, MD, Principal Investigator — Midwest Cardiovascular Research Foundation
Locations (1):
- Trinity Medical Center, Bettendorf, Iowa, United States

REFERENCES:
- [Background] Tepe G, Zeller T, Albrecht T, Heller S, Schwarzwalder U, Beregi JP, Claussen CD, Oldenburg A, Scheller B, Speck U. Local delivery of paclitaxel to inhibit restenosis during angioplasty of the leg. N Engl J Med. 2008 Feb 14;358(7):689-99. doi: 10.1056/NEJMoa0706356. PMID 18272892
- [Background] Werk M, Langner S, Reinkensmeier B, Boettcher HF, Tepe G, Dietz U, Hosten N, Hamm B, Speck U, Ricke J. Inhibition of restenosis in femoropopliteal arteries: paclitaxel-coated versus uncoated balloon: femoral paclitaxel randomized pilot trial. Circulation. 2008 Sep 23;118(13):1358-65. doi: 10.1161/CIRCULATIONAHA.107.735985. Epub 2008 Sep 8. PMID 18779447
- [Background] Hawkins BM, Hennebry TA. Local paclitaxel delivery for treatment of peripheral arterial disease. Circ Cardiovasc Interv. 2011 Jun;4(3):297-302. doi: 10.1161/CIRCINTERVENTIONS.110.961052. Epub 2011 May 3. No abstract available. PMID 21540442
- [Background] Dake MD, Ansel GM, Jaff MR, Ohki T, Saxon RR, Smouse HB, Zeller T, Roubin GS, Burket MW, Khatib Y, Snyder SA, Ragheb AO, White JK, Machan LS; Zilver PTX Investigators. Paclitaxel-eluting stents show superiority to balloon angioplasty and bare metal stents in femoropopliteal disease: twelve-month Zilver PTX randomized study results. Circ Cardiovasc Interv. 2011 Oct 1;4(5):495-504. doi: 10.1161/CIRCINTERVENTIONS.111.962324. Epub 2011 Sep 27. PMID 21953370
- [Background] Speck U, Scheller B, Abramjuk C, Grossmann S, Mahnkopf D, Simon O. Inhibition of restenosis in stented porcine coronary arteries: uptake of Paclitaxel from angiographic contrast media. Invest Radiol. 2004 Mar;39(3):182-6. doi: 10.1097/01.rli.0000116125.96544.64. PMID 15076010
- [Background] Scheller B, Speck U, Schmitt A, Bohm M, Nickenig G. Addition of paclitaxel to contrast media prevents restenosis after coronary stent implantation. J Am Coll Cardiol. 2003 Oct 15;42(8):1415-20. doi: 10.1016/s0735-1097(03)01056-8. PMID 14563585
- [Background] Herdeg C, Gohring-Frischholz K, Haase KK, Geisler T, Zurn C, Hartmann U, Wohrle J, Nusser T, Dippon J, May AE, Gawaz M. Catheter-based delivery of fluid paclitaxel for prevention of restenosis in native coronary artery lesions after stent implantation. Circ Cardiovasc Interv. 2009 Aug;2(4):294-301. doi: 10.1161/CIRCINTERVENTIONS.108.827865.108.827865. Epub 2009 Jul 22. PMID 20031731
- [Background] Margolis J, McDonald J, Heuser R, Klinke P, Waksman R, Virmani R, Desai N, Hilton D. Systemic nanoparticle paclitaxel (nab-paclitaxel) for in-stent restenosis I (SNAPIST-I): a first-in-human safety and dose-finding study. Clin Cardiol. 2007 Apr;30(4):165-70. doi: 10.1002/clc.20066. PMID 17443649